CLINICAL TRIAL: NCT02482714
Title: Life Quality Determinant Assessment of Fibromyalgia Patients Related to Health Devices
Brief Title: Life Quality Determinant Assessment of Fibromyalgia Patients
Acronym: FIBROQUALLIFE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulty
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 6118
Record Dates: First submitted 2015-06-18; First posted 2015-06-26 (Estimated); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Fibromyalgia
Keywords: Quality of Life; Physical Activity
MeSH Terms: conditions — Fibromyalgia; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rehab Institute (Experimental): This group will do some physical activity in a specialized institute
  Interventions: Behavioral: Physical activity.
- Club structure (Active Comparator): This group will do some physical activity in a club.
  Interventions: Behavioral: Physical activity.

INTERVENTIONS:
Behavioral: Physical activity. — Have subject do moderate physical activity.

SUMMARY:
The primary purpose is the evaluation of life quality of Fibromyalgia patients. The investigators' main hypothesis includes the role of geographical, sociological, psychological and physical activity on life quality.

ELIGIBILITY:
Inclusion criteria:

* Age group : 20 to 60
* Male or female
* American College of Rheumatology criteria
* Social Security beneficiary
* Informed consent of the patient
* Patient informed of the medical examination prior to inclusion
* Patient residing in the Bas-Rhin area

Exclusion Criteria:

* No medical objections to performing a stress test
* Any cardio-respiratory and musculoskeletal affection preventing physical activity
* Any particular clinical form disease
* Patient in situation of exclusion
* Subject incapacity to understand informed consent
* Patient deprived of freedom or under the protection of a conservator
* Pregnancy or breast-feeding

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Quality of Life with Fibromyalgia score on questionnary QIF (Quality of Life with Fibromyalgia) | 6th month

SECONDARY OUTCOMES:
Score on questionnary Short Form (36) SF36 | 6th month
Measurement of displacement with Global Positioning System GPS | 6th month

CONTACTS AND LOCATIONS:
Overall Officials: Jehan Lecocq, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- University Hospital, Strasbourg, france, Strasbourg, France